CLINICAL TRIAL: NCT06592339
Title: An Open-Label, Randomized, Single-Dose, 3-Period, Crossover Study to Evaluate the Comparative Bioavailability of MK-0616 Capsules and Tablet Formulations in Healthy Participants
Brief Title: A Study of MK-0616 in Healthy Adult Participants (MK-0616-009)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0616-009; MK-0616-009 (Other: MSD)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — MK-0616

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence 1: MK-0616 Reference capsule→MK-0616 Formulation 1 (F1)→MK-0616 Formulation 2 (F2) (Experimental): Period 1: Participants receive MK-0616 reference capsule single dose on Day 1 orally (Period 1 = 15 days). Period 2: Participants receive MK-0616 F1 single dose on Day 1 orally (Period 2 = 15 days). Period 3: Participants receive MK-0616 F2 single dose on Day 1 orally (Period 3 = 15 days). A washout period of 14 days will separate Period 1, Period 2 and Period 3.
  Interventions: Drug: MK-0616
- Sequence 2: MK-0616 Reference capsule→MK-0616 F2→MK-0616 F1 (Experimental): Period 1: Participants receive MK-0616 reference capsule single dose on Day 1 orally (Period 1 = 15 days). Period 2: Participants receive MK-0616 F2 single dose on Day 1 orally (Period 2 = 15 days). Period 3: Participants receive MK-0616 F1 single dose on Day 1 orally (Period 3 = 15 days). A washout period of 14 days will separate Period 1, Period 2 and Period 3.
  Interventions: Drug: MK-0616
- Sequence 3: MK-0616 F1→MK-0616 Reference capsule→MK-0616 F2 (Experimental): Period 1: Participants receive MK-0616 F1 single dose on Day 1 orally (Period 1 = 15 days). Period 2: Participants receive MK-0616 reference capsule single dose on Day 1 orally (Period 2 = 15 days). Period 3: Participants receive MK-0616 F2 single dose on Day 1 orally (Period 3 = 15 days). A washout period of 14 days will separate Period 1, Period 2 and Period 3.
  Interventions: Drug: MK-0616
- Sequence 4: MK-0616 F1→MK-0616 F2→MK-0616 Reference capsule (Experimental): Period 1: Participants receive MK-0616 F1 single dose on Day 1 orally (Period 1 = 15 days). Period 2: Participants receive MK-0616 F2 single dose on Day 1 orally (Period 2 = 15 days). Period 3: Participants receive MK-0616 reference capsule single dose on Day 1 orally (Period 3 = 15 days). A washout period of 14 days will separate Period 1, Period 2 and Period 3.
  Interventions: Drug: MK-0616
- Sequence 5: MK-0616 F2→MK-0616 Reference capsule →MK-0616 F1 (Experimental): Period 1: Participants receive MK-0616 F2 single dose on Day 1 orally (Period 1 = 15 days). Period 2: Participants receive MK-0616 reference capsule single dose on Day 1 orally (Period 2 = 15 days). Period 3: Participants receive MK-0616 F1 single dose on Day 1 orally (Period 3 = 15 days). A washout period of 14 days will separate Period 1, Period 2 and Period 3.
  Interventions: Drug: MK-0616
- Sequence 6: MK-0616 F2→MK-0616 F1→MK-0616 Reference capsule (Experimental): Period 1: Participants receive MK-0616 F2 single dose on Day 1 orally (Period 1 = 15 days). Period 2: Participants receive MK-0616 F1 single dose on Day 1 orally (Period 2 = 15 days). Period 3: Participants receive MK-0616 reference capsule single dose on Day 1 orally (Period 3 = 15 days). A washout period of 14 days will separate Period 1, Period 2 and Period 3.
  Interventions: Drug: MK-0616

INTERVENTIONS:
Drug: MK-0616 — oral administration

SUMMARY:
The goal of the study is to learn what happens to levels of MK-0616 in the blood when MK-0616 is given in different forms. Researchers believe that there is no effect on a healthy person's body if MK-0616 is given in different forms.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health before randomization
* Has a body mass index (BMI) ≥18 and ≤32 kg/m^2, inclusive

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, GI, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cancer with pre-specified exceptions (adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix or other malignancies that have been successfully treated with appropriate follow up and therefore unlikely to recur for the duration of the study, per protocol guidelines)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of MK-0616 | Predose and at designated timepoints up to 168 hours postdose
  Blood samples will be collected to determine the AUC0-inf of MK-0616.
Area Under the Concentration-Time Curve from Time 0 to 24 hours (AUC0-24hr) of MK-0616 | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the AUC0-24 of MK-0616.
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of MK-0616 | Predose and at designated timepoints up to 168 hours postdose
  Blood samples will be collected to determine the AUC0-last of MK-0616.
Maximum Plasma Concentration (Cmax) of MK-0616 | Predose and at designated timepoints up to 168 hours postdose
  Blood samples will be collected to determine the Cmax of MK-0616.
Maximum Plasma Concentration (C24) of MK-0616 | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the C24 of MK-0616.
Apparent Terminal Half-life (t1/2) of MK-0616 | Predose and at designated timepoints up to 168 hours postdose
  Blood samples will be collected to determine the apparent t1/2 of MK-0616.
Time to Maximum Plasma Concentration (Tmax) of MK-0616 | Predose and at designated timepoints up to 168 hours postdose
  Blood samples will be collected at pre-specified timepoints to determine the Tmax of MK-0616.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 2 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Due to an AE | Up to approximately 2 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- QPS-MRA, LLC-Early Phase, South Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com